CLINICAL TRIAL: NCT06099301
Title: Brief Advice of a List of Mental Health Mobile Apps for Reducing Depressive Symptoms and Anxiety in Adults: a Pilot Randomised Controlled Trial
Brief Title: Mental Health Mobile Apps for Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Dr Grace SUN Yuying, Assistant Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-HMRF2023/09
Record Dates: First submitted 2023-10-16; First posted 2023-10-25 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Depressive Symptoms; Anxiety; Well-Being, Psychological
Keywords: Apps; Depressive Symptoms; Anxiety; Mental Health; Coping Self-efficacy
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Waitlist control (WC) (No Intervention): The WC group will not receive treatment from the research team during the assessment period. But they will be notified their evaluation results (mild to moderate depression) after they complete the baseline assessment. They will receive the information about mental health hotline services for general public (e.g. Social Welfare Department: 2343 2255; Caritas Family Crisis Support Centre: 18288; Joyful Mental Health Foundation: 2301 2303). The intervention group will receive the hotline information as well. If they want to consult a family doctor, information about the primary care provider/directory for mental health care and counselling services will be provided in their preferred district. Their treatment or help-seeking of the formal mental health services will not be intervened. The mobile app list will be provided to the WC group after the assessment period. The instruction session will be delivered to the WC group and provide necessary assistance.
- Brief advice of a list of mobile apps (Experimental): In the instruction session, the participants will be introduced with the concept of self-care, a list of four mobile apps with high quality and suitability, and the main functions of these apps. Participants will be instructed to use at least one of the apps for 10 min each day for 30 days. They have freedom to choose which one app to use, or a mix of two or three apps. For each app they choose, they will create user accounts by themselves but be reminded to protect privacy. Two reminders will be sent to the participants at the 2nd and 3rd week. The message will include reminders to use the suggested mobile apps, self-care concept, and tips of using the provided apps. If they have not accessed to any of the mobile apps, the project coordinator will discuss the reasons and work together with the participants to overcome the problems.
  Interventions: Behavioral: Brief advice of a list of mobile apps

INTERVENTIONS:
Behavioral: Brief advice of a list of mobile apps — The mobile apps in the list should: (1) focus primarily on anxiety/depression/stress, (2) be available for free download; (3) be available in English or Chinese; and (4) have a user star rating in the app store.
  Other Names: mobile apps
  Arms: Brief advice of a list of mobile apps

SUMMARY:
In Hong Kong, the shortage of mental health professionals has been a public health concern for many decades. The World Health Organization (WHO) recommends self-care intervention as one of the most promising and exciting new approaches to improve health and well-being. Rapid development in digital technologies is making population-based self-care interventions possible. The goal of this pilot randomised controlled trial is to provide brief advice of a list of mental health mobile apps for reducing depressive symptoms and anxiety in adults. Participants will be instructed to use four mobile apps for 10 min each day for 30 days. They have freedom to choose which one app to use, or a mix of two or three apps. The Waitlist control group will not receive treatment from the research team during the assessment period. But they will be notified their evaluation results (mild to moderate depression) after they complete the baseline assessment. They will receive the information about mental health hotline services for general public. The hypothesis is that the interventions show preliminary effectiveness in reducing adults' depressive and/or anxiety symptoms.

DETAILED DESCRIPTION:
Over 10,000 mental health mobile apps are commercially available and counting. Only a small number of apps are regularly downloaded and used, which is in stark contrast with the surge of depression and anxiety apps on the marketplace. Most commercial apps were released without any supportive data. It is costly to develop a brand-new app, which requires a professional team to maintain. The reach and impact are questionable. Some apps include rich contents, yet the public or patients may find them not useful. The preferences of mobile apps may vary in different populations. A list of the high-quality mobile apps will be formed, then conduct a pilot randomized controlled trial (RCT) to evaluate whether a brief advice to provide these apps is feasible for adult populations with mild to moderate depressive symptoms. The assumption is that digital-based self-help interventions are effective methods to improve wellbeing and promote mental health, and their impact could be extended at the population level with a minimal cost and time if proved to be effective. In this feasibility trial, the research aim was to explore trial design, subject acceptability of the interventions and preliminary effectiveness of the interventions, and to provide data to estimate the parameters required to design a definitive RCT.

A parallel-group pilot RCT with an equal randomization of 1:1, (1) Intervention group: brief advice of a list of mobile apps (LMA) and (2) Waitlist control (WL) group. A total of 234 participants (117 in each group) who have mild to moderate depression or anxiety symptoms will be recruited. Participants will be approached through mass email, public posters or active approach in community centres. The randomisation will be conducted after the participants give consent and complete the baseline assessments (T1) (via Qualtrics). The individuals will be randomised into intervention and control groups. The randomized list will be generated using an Excel spreadsheet by a statistician who is not involved in any part of the study. The recruitment staff will be blinded in the allocation process. The randomisation number will not be decoded to the participants until they get assigned a group. Considering the nature of the intervention, participants and research staff cannot be blinded in the process. As the recruitment will be mainly conducted online and through telephone, contamination between groups is expected to be minimal. Potential contamination will be checked at the T1 assessment by asking whether any participants they know have attended the other group. In the final assessment, the participants in the control group will be asked whether they have used any of the recommended apps in the past 3 months.

A 2-hour instruction session of the mobile apps will be delivered to all the participants via Zoom or other online platforms. Participants will be introduced to the concept of self-care and presented with a list of four high-quality and suitable mobile apps along with their main functions. Participants will be instructed to use at least one of the apps for 10 minutes daily over a period of 30 days. They can choose one app or a combination of two or three apps. Participants will create their own user accounts for the chosen app(s), with a reminder to prioritize privacy. Two reminders will be sent during the second and third weeks, emphasizing app usage, the concept of self-care, and providing tips for using the apps. If participants encounter any difficulties accessing the apps, the project coordinator will discuss the issues and collaborate with them to find solutions. Participants will complete the process evaluation (intervention group only) immediately after the intervention (T2), complete the process evaluation (intervention group only) and outcome assessment at 3-month (T3). A fidelity checks on adherence and competence will be conducted.

The feasibility outcomes, including the recruitment rate and duration, retention rate, and adverse events, will be reported descriptively and narratively. For the clinical endpoints, descriptive statistics, mean (standard deviation) for continuous outcomes, will be reported. After adjusting the baseline covariates, mean differences in the outcomes will be compared between the two groups. Multiple imputation approach will be used to deal with missing data (mice package in R). Three sensitivity analyses will be carried out to assess the effect of three factors on the outcomes (retention, choice of mobile apps, effective features). For the in-depth telephone interview, content analysis method will be used following the framework method analysis procedure (e.g., coding). It is expected that the intervention group show more significant improvements in the measured outcomes than the control group, indicating preliminary evidence of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* Have mild to moderate depression (Patient Health Questionnaire (PHQ) - 9, score 5-14) and/or anxiety (General Anxiety Disorder (GAD) - 7, score 5-14)
* Hong Kong residents who can communicate in Chinese (Cantonese)
* Own a smart phone

Exclusion Criteria:

* Physically or mentally unable to communicate
* Currently taking antidepressant or anxiolytic medication or receiving active psychotherapy in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in depressive symptoms | T1: baseline; T2: immediate post-intervention (1-month after baseline); T3: 3-month after the intervention
  The Patient Health Questionnaire (PHQ)-9 will be used to measure depressive symptoms. Participants rate the frequency of nine symptoms over the past two weeks on a 4-point Likert scale (from 0=not at all to 3=nearly every day). The total score ranges from 0 to 27, with higher scores indicating a greater severity of depressive symptoms.
Changes in anxiety symptoms | T1: baseline; T2: immediate post-intervention (1-month after baseline); T3: 3-month after the intervention
  The Generalized Anxiety Disorder (GAD)-7 will be used to measure anxiety symptoms. Participants rate the frequency of seven symptoms over the past two weeks on a 4-point Likert scale (from 0=not at all to 3=nearly every day). The total score ranges from 0 to 21, with a higher score indicating a higher level of anxiety.

SECONDARY OUTCOMES:
Changes in well-being | T1: baseline; T2: immediate post-intervention (1-month after baseline); T3: 3-month after the intervention
  The 7-item Short Warwick-Edinburgh Mental Well-being Scale with the 5-point Likert scale (1=none of the time, 5=all the time) will be used to measure well-being. The score is calculated by summing all seven items with a range of 7 to 35. A higher score indicates a higher level of well-being.
Changes in coping self-efficacy (CSE) | T1: baseline; T2: immediate post-intervention (1-month after baseline); T3: 3-month after the intervention
  The Coping Efficacy Questionnaire (CEQ) with the 4-point Likert scale (1 = totally disagree, 4 = strongly agree) will be used to assess CSE. Scores are calculated from the sum of the reverse score of items 1-3, and the remaining 4-17 item scores, ranging from 17 to 68. Higher scores indicate greater CSE.
Changes in psychological stress | T1: baseline; T2: immediate post-intervention (1-month after baseline); T3: 3-month after the intervention
  The Chinese version of the Perceived Stress Scale-10 (CPSS-10) will be used to measure psychological stress during the past month. It consists of six positive and four negative items, with each item scored on a 5-point Likert scale from 0 (never) to 4 (very often). The positive items will be reverse scored. The total score ranges from 0 to 40, and a higher score indicates a higher perceived psychological stress.

OTHER OUTCOMES:
Utility assessment during application use | T2: immediate post-intervention (1-month after baseline); T3: 3-month after the intervention
  At T2 and T3, participants in the intervention group will report the mobile app they have used (multiple choices of 3 apps), perceived usefulness of the app (0-10, with "0" indicating "not useful at all" and "10" indicating "very useful"), satisfaction of the apps (level of satisfaction: 0-10, with "0" indicating "unsatisfied" and "10" indicating "satisfied"), perceived need of using formal mental health services (0-10, with "0" indicating "no need at all" and "10" indicating "much needed"), subjective changes in personal mental health and wellbeing (1-5, with "1" indicating "much worse" and "5" indicating "much better").
The overall satisfaction with the program and subjective changes | After completing all quantitative outcome assessments (3-month after the intervention)
  In-depth telephone interviews will be conducted with 30 subjects in the intervention group (15 participants who used the apps at least once in the 3-4th week reported at T2 & 15 participants who did not use the apps in the 3-4th week). Each interview will last around 15 minutes. The interviews will explore subjects' satisfaction with the program content, subjective changes, factors, process or reasons for the subjective changes, difficulties in practice, barriers in using the apps in daily life, and suggestions for selection of the apps and future programs. The project coordinator will serve as a moderator in the interviews. All interviews will be audio-recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Sun, PhD, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hong Kong